CLINICAL TRIAL: NCT04266106
Title: Effect of Perioperative Probiotics on Clinical Outcomes of Patients Undergoing Major Abdominal Operation in Community Settings - 2
Brief Title: Probiotics and Recovery From Gastrointestinal Surgery - 2
Acronym: PROGRESS-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jan Franko, MD (Other)
Collaborators: SuperBio (Unknown)
Responsible Party: Sponsor-Investigator, Jan Franko, MD, Chair of Surgical Oncology, MercyOne Des Moines Medical Center
Organization: MercyOne Des Moines Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MMC-2019-56
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Surgical Recovery

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo
- probiotic (Experimental)
  Interventions: Drug: SuperBio probiotic

INTERVENTIONS:
Drug: SuperBio probiotic — One capsule po BID for 28 days
  Arms: probiotic
Drug: Placebo — One capsule po BID for 28 days
  Arms: Placebo Comparator

SUMMARY:
This prospective randomized trial is designed to test a pragmatic simple intervention in a community hospital. The trial will test the hypothesis whether patient recovery after a major elective abdominal operation can be improved and/or accelerated with postoperative use of probiotics.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years undergoing elective major abdominal operation
* Functional GI tract expected after operation

Exclusion Criteria:

* Current episode of acute necrotizing pancreatitis as defined by surgeon
* Palliative decompressive GI tube
* Life expectancy ≤ 6 months
* Systemic immune-mediated disease active requiring systemic therapy:
* Prednisone ≥20 mg QD
* IV immunoglobulins
* Anti-rejection medication
* Presence of functional transplanted organ
* Systemic collagen-related disease treated with immunomodulating agents, including rheumatoid arthritis, SLE, scleroderma, etc.
* Topical chemotherapy or corticosteroids, and chemotherapy applied during operation are allowed
* Patient taking probiotics, synbiotics, or cobiotics as part of their lifestyle
* Need for full systemic anticoagulation postoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | up to 2 months
  Functional Assessment of Cancer Therapy (FACT) G7 score: higher value corresponds with better QoL, range 0-28 points

CONTACTS AND LOCATIONS:
Overall Officials: Jan Franko, Principal Investigator — MercyOne Des Moines Medical Center
Locations (1):
- MercyOne Des Moines Medical Center, Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
No sharing

REFERENCES:
- [Background] Franko J, Raman S, Krishnan N, Frankova D, Tee MC, Brahmbhatt R, Goldman CD, Weigel RJ. Randomized Trial of Perioperative Probiotics Among Patients Undergoing Major Abdominal Operation. J Am Coll Surg. 2019 Dec;229(6):533-540.e1. doi: 10.1016/j.jamcollsurg.2019.09.002. Epub 2019 Sep 25. PMID 31562911